CLINICAL TRIAL: NCT03170908
Title: Pragmatic Strategies for Assessing and Enhancing High Fidelity Delivery of Interpersonal Psychotherapy (IPT) in Community Practice
Brief Title: Effective Implementation of Interpersonal Psychotherapy
Status: Terminated | Type: Observational
Why Stopped: Conflict of Interest (COI) cannot be managed
Sponsor: University of Iowa (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 201705766; 1R01MH112624 (NIH)
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase I Patients: Patients with depression receiving community-based services will receive Interpersonal Psychotherapy
  Interventions: Behavioral: Interpersonal Psychotherapy
- Phase II Patients: Patients with depression receiving community-based services will receive Interpersonal Psychotherapy
  Interventions: Behavioral: Interpersonal Psychotherapy

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy — Interpersonal Psychotherapy (IPT) is an empirically-validated time-limited treatment for depression

SUMMARY:
The study is designed to observe the impact of improved measures of the fidelity on the community delivery of Interpersonal Psychotherapy. Pairs of therapist-patient dyads will be observed, first to develop and test brief measures of fidelity, and then to correlate those measures with symptomatic outcomes.

DETAILED DESCRIPTION:
The study is designed to observe the impact of improved measures of the fidelity on the community delivery of Interpersonal Psychotherapy. In Phase I, 250 pairs of therapist-patient dyads will be observed as IPT Fidelity measures are developed and validated. In Phase II, 175 pairs of therapist-patient dyads will be observed to prospectively validate the IPT Fidelity measures with longitudinal outcomes on the PHQ-9.

ELIGIBILITY:
Inclusion Criteria:

* age 18-99
* diagnosis of depressive disorder
* being treated with IPT in community settings

Exclusion Criteria:

- none

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-99 seeking psychotherapy for depression in community-based agencies
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
PHQ-9 | one year
  Patient Health Questionnaire-9

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
we do not plan to share IPD